CLINICAL TRIAL: NCT03576807
Title: The Clinical Research of Anti-CD20 CAR-T Cells in Patients With Refractory or Relapsed B Lymphocyte Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xin Wang (Other)
Responsible Party: Sponsor-Investigator, Xin Wang, The clinical research of targeted CD20-CART cells treatment for refractory or recurrence B lymphocyte lymphoma, Shanghai Longyao Biotechnology Inc., Ltd.
Organization: Shanghai Longyao Biotechnology Inc., Ltd. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHLY1701
Record Dates: First submitted 2018-06-21; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-04

CONDITIONS: Relapsed or Refractory B-cell Lymphomas
Keywords: B-cell leukemia
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD20 CAR-T cells (Experimental): Experimental: CD20 CAR-T cells
  Interventions: Drug: CD20 CAR-T cells

INTERVENTIONS:
Drug: CD20 CAR-T cells — A total of 1 - 20×10^6 CD20 CAR-T cells/kg will be administered by IV infusions.

SUMMARY:
The present study is an exploratory study. Patients who meeting the enrollment conditions for relapsed or refractory B-cell lymphoma receive a single intravenous dose of CD20-CART cells. The research with the open-label, single arm running control methods in order to initially observe the safety, tolerability, and cellular pharmacokinetics of CD20-CART cell drugs.

DETAILED DESCRIPTION:
The main purpose:

To preliminary explore the safety, tolerability and cellular pharmacokinetics of CD20-CART cell agents in the treatment of relapsed or refractory B-cell lymphomas.

The Secondary purpose:

The following indicators for preliminary observations of CD20-CART cells in the treatment of relapsed or refractory B-cell malignant lymphoma.

1. The determination of lymph nodes to evaluate the anti-tumor effect caused by the input of CD20-CART cells agents.
2. Assessing the ability of CD20-CART cell agents to inhibit the migration of bone marrow and lymph node tumor foci.
3. Assess the killing ability of CD20-CART cell agents to tumor cells in vitro, for patients whose tumor cells could obtain.
4. Disease control rate (DCR) (=CR (complete disease remission) + PR (partial remission of disease) + SD (stable disease), short-term efficacy assessment); Overall survival (OS) and progression-free survival (PFS) (long-term efficacy assessment).

ELIGIBILITY:
Inclusion Criteria:

1．Patients diagnosed with B-cell relapse/refractory lymphoma have no effective treatment option. They have been treated for more than 2 years after autologous or allogeneic stem cell transplantation.

2.The patient's age is between 10 and 80 years old. 3. The expected survival of the patient is greater than 12 weeks. 4. Important organ functions must meet the following conditions: The echocardiography indicates that the cardiac ejection fraction is ≥50%. Electrocardiogram showed no obvious abnormalities. Creatinine clearance was calculated using the Cockcroft-Gault formula ≥ 40 ml/min. ALT value and AST value ≤ 3 times normal range. Total bilirubin ≤2.0mg/dl. The coagulation function showed a PT value and APPT value less than 2 times normal. Arterial oxygen saturation (SpO2) is greater than 92%.

5. Blood routine parameters: Hgb≥80g/L, ANC≥1×109/L, PLT≥50×109/L. 6. The pregnancy test for women of childbearing age must be negative; both male and female patients must agree to use effective contraceptives during the treatment period and within the next year; 7. There are measurable target lesions, see annex to measure lesion definition. 8. Patients have sufficient venous access to apheresis or venous blood and no other leukocyte isolation contraindications.

9.ECOG评分≤2. 10. Patients need to sign informed consent.

Exclusion Criteria:

1. The patient is a pregnant or breastfeeding woman, or is a woman with a pregnancy plan within six months;
2. Patients have infectious diseases (such as HIV, RPR, active tuberculosis, etc.);
3. The patient is an active hepatitis B or hepatitis C infection.
4. The patient received genetic product treatment within six months.
5. The patient participated in a clinical trial within six months.
6. The patient has a severe autoimmune disease.
7. The doctor thinks that there are other reasons that can't be accepted.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-04-03 (Estimated); Study Completion 2020-04-03 (Estimated)

PRIMARY OUTCOMES:
Study related adverse events [ Time Frame: 4 weeks ] | 4 weeks
  Occurrence of study related adverse events, defined as NCI CTC ≥ Grade 3 signs/symptoms, laboratory toxicities and clinical events that are possible.

SECONDARY OUTCOMES:
Graft Activity Endpoint Detection | 24 hours, 1 week, 2 weeks, 3 weeks, 4 weeks, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 1 quarter, 2 quarters, 3 months after returning to CART cells. Data were collected in quarters, 4 quarters, 5 quarters, 6 quart
  The PCR method was used to detect the copy number of the exogenous CAR vector in the blood until the end of the test was negative for both tests.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided